CLINICAL TRIAL: NCT04499079
Title: Alliances to Disseminate Addiction Prevention and Treatment (ADAPT): A Statewide Learning Health System to Reduce Substance Use Among Justice-Involved Youth in Rural Communities
Brief Title: Alliances to Disseminate Addiction Prevention and Treatment (ADAPT)
Acronym: ADAPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Matthew Aalsma, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1910282231; UG1DA050070 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Substance-Related Disorders; Recidivism; Opioid-Related Disorders; Substance Use; Criminal Behavior
Keywords: Juvenile Justice Behavioral Health Services Cascade
MeSH Terms: conditions — Substance-Related Disorders; Recidivism; Opioid-Related Disorders; Criminal Behavior | interventions — Learning Health System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probation Referral Practice as Usual (No Intervention): Data are collected regarding standard probation practice and outcomes before implementation of the Learning Health System.
- Learning Health System (Experimental): Participating counties receive a system-level intervention, a Learning Health System, designed to improve youth connection to substance use treatment.
  Interventions: Other: Learning Health System

INTERVENTIONS:
Other: Learning Health System — This is a system-level intervention designed to improve collaboration among personnel from the juvenile and behavioral healthcare systems.
  Arms: Learning Health System

SUMMARY:
Youth involved in the juvenile justice system (YJJ) bear a disproportionate burden of the addiction crisis. YJJ substance use (SU) is extremely prevalent, with a third of YJJ meeting criteria for a substance use disorder (SUD). The investigators seek to address the national addiction crisis at its epicenter.

Despite their high need for SUD services, and the proliferation of evidence-based interventions to reduce SU, YJJ are rarely connected to needed, high-quality SU care. A care cascade model highlights gaps in YJJ achieving the full continuum of SUD care (i.e., SUD risk identification, treatment referral, treatment initiation, and treatment engagement). YJJ on community supervision/probation face a unique problem accessing SUD services; while the courts or probation may identify YJJ need for SUD care, YJJ must receive care through healthcare agencies in the community. The primary goal of the project, Alliances to Disseminate Addiction Prevention and Treatment (ADAPT) is to address this and other gaps along the care cascade for YJJ. The investigators will accomplish this goal by creating alliances between the juvenile justice system (JJ) agencies and community mental health centers (CMHCs) in eight Indiana counties.

ADAPT takes a two-pronged approach. First, the investigators will employ a Learning Health System (LHS) to develop collaborative alliances between JJ agencies and CMHCs, organizations that traditionally operate independently. Second, the investigators will present local Cascade data during continuous quality improvement cycles within the LHS alliances. By offering agency representatives an opportunity to view and discuss, for example, the local rate at which YJJ with SUD risk are initiating CMHC SU services, the investigators will facilitate development of tailored, local solutions to improve the Cascade for each county's YJJ.

To maximize long-term sustainability of ADAPT's JJ-CMHC alliances, the investigators will conduct this research in collaboration with leaders from an existing statewide initiative, the Juvenile Detention Alternatives Initiative (JDAI). JDAI is a juvenile justice reform effort that utilizes data-driven decision-making and is implemented in almost 300 counties across the US. If this project is successful, the JDAI infrastructure and support for this research will inform sustainment and expansion across Indiana and the nation.

The investigators hypothesize that ADAPT - novel LHS alliances using Cascade data to implement localized solutions to YJJ receiving evidence-based addictions care - will positively impact SU and recidivism outcomes over time. The investigators seek to complete the following specific aims:

AIM 1: Implement LHS alliances between JJ agencies and CMHCs. The investigators will establish LHS alliances: novel, collaborative partnerships between JJ agencies and CMHCs.

AIM 2: Generate and track local solutions to address gaps in the Cascade for YJJ in rural Indiana counties. Quantifying local Cascade data will enable JJ agencies and CMHCs to suggest and implement tailored, evidenced-based interventions, which will be tracked through LHS quality improvement cycles.

AIM 3: Assess implementation outcomes and processes. We will assess implementation outcomes, such as system alliance, among JJ and CHMC personnel using mixed methods.

AIM 4: Assess the impact of ADAPT. Conduct a stepped wedge cluster randomized controlled trial to assess the impact of LHS alliances on the Cascade for YJJ. We will analyze administrative data linked across JJ and health systems to assess the long-term, community-wide effects of ADAPT on public health and safety outcomes (e.g., lower rates of SU-related outcomes and criminal recidivism).

ELIGIBILITY:
Youth Inclusion Criteria:

* Reside in a participating county assigned to receive the LHS intervention
* Utilized any local CMHC service during the 24-month intervention period
* Age 11 to 22 years old

Youth Exclusion Criteria:

* N/A

Ages: 11 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12400 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Utilization of substance use treatment services | 10 years
  Completion of substance use treatment, completion of substance use classes, enrollment in medication assisted treatment
Recidivism | 10 years
  Rate of re-offense
Substance use related health outcomes | 10 years
  Hospital and emergency department visits related to substance use

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aalsma MC, Schwartz K, Sun D, O'Reilly LM, Brown SA, Monahan PO, Saldana L, Wiehe SE, Zapolski TCB, Hulvershorn LA, Adams ZW, Dir AL. Learning Health Systems and Substance Use Care Cascade Achievement Among Justice-Involved Youth: A Cluster-Randomized Stepped-Wedge Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2558222. doi: 10.1001/jamanetworkopen.2025.58222. PMID 41665903
- [Derived] O'Reilly L, Sun D, Schwartz K, Gillenwater L, Dir A, Monahan P, Aarons GA, Saldana L, Adams Z, Zapolski T, Hulvershorn L, Aalsma MC. Impact of learning health systems on cross-system collaboration between youth legal and community mental health systems: a type II hybrid effectiveness-implementation trial. Implement Sci Commun. 2024 Dec 24;5(1):142. doi: 10.1186/s43058-024-00686-6. PMID 39719625
- [Derived] Ahrens K, Blackburn N, Aalsma M, Haggerty K, Kelleher K, Knight DK, Joseph E, Mulford C, Ryle T, Tolou-Shams M. Prevention of Opioid Use and Disorder Among Youth Involved in the Legal System: Innovation and Implementation of Four Studies Funded by the NIDA HEAL Initiative. Prev Sci. 2023 Oct;24(Suppl 1):99-110. doi: 10.1007/s11121-023-01566-6. Epub 2023 Jul 1. PMID 37393415